CLINICAL TRIAL: NCT01802125
Title: Observational - SNP Array Analysis of Undifferentiated Sarcomas
Brief Title: Biomarker Differences in Samples From Patients With Undifferentiated Sarcomas
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST12B9; NCI-2013-00489 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Basic science (SNP array analysis): Tissue samples are analyzed using laboratory biomarker analysis for LOH and SNP array profiling using microarray and immunohistochemistry.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies biomarker differences in samples from patients with undifferentiated sarcomas. Studying biomarker in tissue samples from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer

DETAILED DESCRIPTION:
Study Subtype: Ancillary/Correlative Observational Study Model: Cohort Time Perspective: Prospective Biospecimen Retention: Samples With DNA Biospecimen Description: Tissue Study Population Description: Patients from ARST0332 study Sampling Method: Non-Probability Sample

PRIMARY OBJECTIVES:

I. To determine what proportion of unclassifiable sarcomas are unclassifiable because the initial evaluation was not sufficiently comprehensive versus what proportion can be regarded as "true" undifferentiated sarcoma when a comprehensive assessment has been performed.

II. To develop formal diagnostic criteria for establishing the diagnosis of undifferentiated sarcoma.

III. To determine whether undifferentiated sarcoma can be subdivided into separate and distinct pathologic entities that are distinguishable by light microscopy, immunohistochemistry, single nucleotide polymorphism (SNP) array profiling, or clinical features.

IV. To determine whether undifferentiated sarcomas with specific "actionable mutations" can be identified based on their histologic appearance, immunohistochemical staining characteristics, or SNP array profiling features.

OUTLINE:

Tissue samples are analyzed for loss of heterozygosity (LOH) and SNP array profiling using microarray and immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* 49 cases of undifferentiated sarcomas from ARST0332 (additional cases may be ascertained as eligible for this current project that also fall under ARST0332 to be requested later if necessary)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Undifferentiated sarcomas from ARST0332
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Proportion of unclassifiable sarcomas that are unclassifiable | Baseline
Development of formal diagnostic criteria for establishing the diagnosis of undifferentiated sarcoma | Baseline
Separate and distinct pathologic entities of undifferentiated sarcoma that are distinguishable by light microscopy, immunohistochemistry, SNP array profiling, or clinical features | Baseline
Specific "actionable mutations" that can be identified based on their histologic appearance, immunohistochemical staining characteristics, or SNP array profiling features | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Julia Bridge, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States